CLINICAL TRIAL: NCT01407822
Title: A National, Multi Center, Randomized, Open-label, Phase II Trial of Erlotinib Versus Combination of GC as (Neo)Adjuvant Treatment in Stage IIIA-N2 NSCLC With Sensitizing EGFR Mutation in Exon 19 or 21(EMERGING)
Brief Title: Erlotinib Versus Gemcitabine/Cisplatin as (Neo)Adjuvant Treatment in Non-small Cell Lung Cancer
Acronym: EMERGING
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Guangdong Association of Clinical Trials (Other)
Collaborators: Guangdong Provincial People's Hospital (Other); Tianjin Medical University Cancer Institute and Hospital (Other); Jilin Provincial Tumor Hospital (Other); Jiangsu Cancer Institute & Hospital (Other); Zhejiang Cancer Hospital (Other); Peking University Cancer Hospital & Institute (Other); Sun Yat-sen University (Other); West China Hospital (Other); The First Affiliated Hospital of Dalian Medical University (Other); Peking University People's Hospital (Other); Xi'an Jiaotong University (Other); Shanghai Zhongshan Hospital (Other); Guangzhou General Hospital of Guangzhou Military Command (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); Fujian Medical University Union Hospital (Other); Linyi Tumour Hospital (Other); Northern Jiangsu People's Hospital (Other)
Responsible Party: Principal Investigator, Yi-Long Wu, Dr, Guangdong Association of Clinical Trials
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTONG 1103; ML25304 (Other Grant/Funding Number: Roche); NCT01392404 (obsolete NCT alias)
Record Dates: First submitted 2011-07-26; First posted 2011-08-02 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Lung cancer; IIIA-N2; Neo-adjuvant treatment; EGFR mutations; Tyrosine kinase inhibitor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Erlotinib Hydrochloride; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Erlotinib arm (Experimental): In the neo-adjuvant treatment phase, erlotinib 150 mg/day taken orally for 6 weeks(42 days).In the post-surgery phase, erlotinib 150mg/day taken orally for 1 year or till disease progression or unacceptable toxicity.
  Interventions: Drug: Erlotinib
- Chemo arm (Active Comparator): In the neo-adjuvant treatment phase, patient will receive gemcitabine 1250mg/m2 IV on day 1 and day 8, and cisplatin 75mg/m2 on day 1 of a 3-week schedule for 2 cycles. In the post-surgery phase, Gemcitabine 1250mg/m2 IV on day 1 and day 8, and cisplatin 75mg/m2 on day 1 of a 3-week schedule for 2 cycles or till disease progression or unacceptable toxicity.
  Interventions: Drug: Gemcitabine/cisplatin

INTERVENTIONS:
Drug: Erlotinib — In the neo-adjuvant treatment phase, erlotinib 150 mg/day taken orally for 6 weeks(42 days).In the post-surgery phase, erlotinib 150mg/day taken orally for 1 year or till disease progression or unacceptable toxicity.
  Other Names: Tarceva
  Arms: Erlotinib arm
Drug: Gemcitabine/cisplatin — In the neo-adjuvant treatment phase, patient will receive gemcitabine 1250mg/m2 IV on day 1 and day 8, and cisplatin 75mg/m2 on day 1 of a 3-week schedule for 2 cycles. In the post-surgery phase, Gemcitabine 1250mg/m2 IV on day 1 and day 8, and cisplatin 75mg/m2 on day 1 of a 3-week schedule for 2 cycles or till disease progression or unacceptable toxicity.
  Other Names: Gemzar/cisplatin
  Arms: Chemo arm

SUMMARY:
Stage IIIA NSCLC represents a relatively heterogeneous group of pts with ipsilateral mediastinal (N2) lymph node involvement. The relative roles of treatment modalities are not clearly defined. Concurrent chemoradiation therapy remains an important treatment for stage IIIA disease, but its treatment-related life threatening toxicity limits its use. The EGFR tyrosine kinase inhibitor (TKI) may provide a dramatic response in pts with pulmonary adenocarcinoma carrying EGFR activating mutations in the metastatic setting. In the OPTIMAL study, first-line erlotinib versus carboplatin/GEM in advanced NSCLC pts with EGFR activating mutations, the primary analysis showed significantly prolonged progressive free survival (PFS) was with erlotinib vs carboplatin/GEM (p<0.0001). The aim of this study is to investigate the efficacy and safety of erlotinib versus GEM plus cisplatin (GC) as neoadjuvant treatment in pts with stage IIIA-N2 NSCLC with EGFR activating mutations and to explore a new treatment strategy for this subset.

DETAILED DESCRIPTION:
Concurrent Chemoradiation therapy remain the standard treatment for stage IIIA disease, but its treatment-related life threaten toxicity limit its use for those pts.

Tarceva monotherapy have been demonstrated a significant improvement in overall survival and disease progression free survival when used for the treatment of patients with metastatic NSCLC, after failure of at least one prior chemotherapy regimen. It is well tolerated without the side effects usually associated with chemotherapy.

Based on the encouraging results reported from the SLCG phase II study reported the efficacy of Tarceva as first line treatment for metastatic NSCLC with EGFR mutation patients would prolong overall survival, delay disease progression and be well tolerated, mOS reached 27 months, ORR reached 71%. Besides, with different mechanism and more tolerable than chemo, Tarceva may provide an important treatment alternative for local advanced pts with EGFR mutation.

In IPASS study (gefitinib or carboplatin/paclitaxel in pulmonary adenocarcinoma as first line treatment), the subgroup of 261 patients who were positive for the epidermal growth factor receptor gene (EGFR) mutation, progression-free survival was significantly longer among those who received gefitinib than among those who received carboplatin-paclitaxel (hazard ratio for progression or death, 0.48; 95% CI, 0.36 to 0.64; P<0.001).

In OPTIMAL study (first-line erlotinib versus carboplatin/gemcitabine in Chinese advanced NSCLC patients with EGFR activating mutations), the primary analysis showed PFS was significantly prolonged with erlotinib vs carboplatin/paclitaxel(13.1months vs 4.6 months, HR 0.16 ; p<0.0001). The objective response rate was significantly improved with erlotinib vs carboplatin/paclitaxel (83% vs 36%, p=0.0000), as was the disease control rate (CR + PR + SD; 96 vs 82%; p=0.002).

The aim of this study is to investigate the efficacy and safety of Tarceva versus combination of Gemcitabine plus Cisplatin as neoadjuvant treatment in patients with stage IIIA- N2 NSCLC with EGFR activating mutation in exon 19 or 21.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent provided.
* Males or females aged ≥18 years.
* Able to comply with the required protocol and follow-up procedures, and able to receive oral medications.
* Pathologically diagnosed of non-small cell lung cancer.
* Diagnosed as stage IIIA- N2.The diagnosis standard of N2 is as below: Pts with resectable stage IIIA-N2 NSCLC confirmed by mediastinoscopy or EBUS or PET/CT.
* EGFR activating mutation in exon 19 or 21 by the biopsy of primary tumor or N2 lymph node.
* Measurable disease must be characterized according to RECIST 1.1 criteria.
* Measurable lesions are defined as those that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 10mm by spiral CT or MRI scan. The measurable criteria of lymph node is the short axis ≥ 15 mm.
* ECOG performance status 0-1.
* Life expectancy ≥12 weeks.
* Adequate hematological function:Absolute neutrophil count (ANC) ≥1.5 x 109/L, and Platelet count ≥100 x 109/L, and Hemoglobin ≥9 g/dL (may be transfused to maintain or exceed this level).
* Adequate liver function: Total bilirubin ≤ 1.5 x upper limit of normal (ULN);Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5 x ULN in subjects without liver metastases; ≤ 5 x ULN in subjects with liver metastases.
* Adequate renal function:Serum creatinine ≤ 1.25 x ULN, and creatinine clearance ≥ 60 ml/min.
* Female subjects should not be pregnant or breast-feeding.

Exclusion Criteria:

* Patients with prior exposure to agents directed at the HER axis (e.g. erlotinib, gefitinib, cetuximab, trastuzumab).
* Patients with prior chemotherapy or therapy with systemic anti-tumour therapy (e.g. monoclonal antibody therapy).
* Resection of primary malignancy.
* EGFR mutation (exon 19 or 21) negative or unknown.
* Uncontrolled central nervous system (CNS) metastasis.
* History of another malignancy in the last 5 years with the exception of the following:Other malignancies cured by surgery alone and having a continuous disease-free interval of 5 years are permitted; Cured basal cell carcinoma of the skin and cured in situ carcinoma of the uterine cervix are permitted.
* Any unstable systemic disease (including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction within the previous year, serious cardiac arrhythmia requiring medication, hepatic, renal, or metabolic disease).
* Known hypersensitivity to Tarceva or gemcitabine or cisplatin.
* Eye inflammation or eye infection not fully treated or conditions predisposing the subject to this.
* Evidence of any other disease, neurological or metabolic dysfunction, physical examination or laboratory finding giving reasonable suspicion of a disease or condition that contraindicated the use of an investigational drug or puts the subject at high risk for treatment-related complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-12-05 (Actual); Primary Completion 2018-04-24 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
The objective response rate (ORR) in neoadjuvant treatment | Tumor response will be evaluated after 6 weeks of induction treatment (during day 43 to day 49).
  To evaluate objective response rate (ORR) of Erlotinib versus combination of Gemcitabine plus Cisplatin as neoadjuvant treatment for stage IIIA- N2 NSCLC with EGFR activating mutation in exon 19 or 21.

SECONDARY OUTCOMES:
Complete resection rate | The patients considered to be technically resectable will undergo resection. Lymph node downstage rate is depended on the pathology dignosis after surgery, an expected average of 8 weeks from randomization.
  To evaluate radical resection rate of two groups.
Pathological complete response (pCR) rate | The patients considered to be technically resectable will undergo resection. Lymph node downstage rate is depended on the pathology dignosis after surgery, an expected average of 8 weeks from randomization.
  To evaluate the pathological complete response (pCR) rate of two groups.
Progression free survival（PFS） | Pts after surgery will receive long-term follow-up including chest CT scan, abdominal ultrasound every 3 months, brain MRI every 6 months, bone scan (ECT) every 12 months for up to 2 years.
  To evaluate Progressive Free Survival (PFS) of two groups.
3 year overall survival (OS) rate | Pts after surgery will receive long-term follow-up including chest CT scan, abdominal ultrasound every 3 months, brain MRI every 6 months, bone scan (ECT) every 12 months for up to 2 years.
  To evaluate the 3 year overall survival (OS) rate of two groups.The third year after surgery is survival follow-up.
Number of Participants with Adverse Events | During the neoadjuvant and adjuvant period, an expected average of 1 years from randomization.
  To evaluate the safety profile(Number of Participants with Adverse Events) of two group.
Quality of Life (QOL) | During the neo-adjuvant treatment phase(1-42 days), surgery treatment phase and adjuvant phase, , an expected average of 1 years from randomization.
  To evaluate the Quality of Life (QOL) of two group

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Long WU, MD, Principal Investigator — Guangdong Lung Cancer Institute; Xue-Ning YANG, MD, Study Chair — Guangdong Provincial People's Hospital; Wen-Zhao ZHONG, MD, Study Director — Guangdong Lung Cancer Institute
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kappers I, Klomp HM, Burgers JA, Van Zandwijk N, Haas RL, van Pel R. Neoadjuvant (induction) erlotinib response in stage IIIA non-small-cell lung cancer. J Clin Oncol. 2008 Sep 1;26(25):4205-7. doi: 10.1200/JCO.2008.16.3709. No abstract available. PMID 18757336
- [Background] Takamochi K, Suzuki K, Sugimura H, Funai K, Mori H, Bashar AH, Kazui T. Surgical resection after gefitinib treatment in patients with lung adenocarcinoma harboring epidermal growth factor receptor gene mutation. Lung Cancer. 2007 Oct;58(1):149-55. doi: 10.1016/j.lungcan.2007.04.016. Epub 2007 Jun 4. PMID 17548126
- [Background] Haura EB, Sommers E, Song L, Chiappori A, Becker A. A pilot study of preoperative gefitinib for early-stage lung cancer to assess intratumor drug concentration and pathways mediating primary resistance. J Thorac Oncol. 2010 Nov;5(11):1806-14. doi: 10.1097/JTO.0b013e3181f38f70. PMID 20881637
- [Background] Rizvi NA, Rusch V, Pao W, Chaft JE, Ladanyi M, Miller VA, Krug LM, Azzoli CG, Bains M, Downey R, Flores R, Park B, Singh B, Zakowski M, Heelan RT, Shen R, Kris MG. Molecular characteristics predict clinical outcomes: prospective trial correlating response to the EGFR tyrosine kinase inhibitor gefitinib with the presence of sensitizing mutations in the tyrosine binding domain of the EGFR gene. Clin Cancer Res. 2011 May 15;17(10):3500-6. doi: 10.1158/1078-0432.CCR-10-2102. Epub 2011 May 10. PMID 21558399
- [Derived] Zhong WZ, Yan HH, Chen KN, Chen C, Gu CD, Wang J, Yang XN, Mao WM, Wang Q, Qiao GB, Cheng Y, Xu L, Wang CL, Chen MW, Kang XZ, Yan WP, Liao RQ, Yang JJ, Zhang XC, Liu SY, Zhou Q, Wu YL. Erlotinib versus gemcitabine plus cisplatin as neoadjuvant treatment of stage IIIA-N2 EGFR-mutant non-small-cell lung cancer: final overall survival analysis of the EMERGING-CTONG 1103 randomised phase II trial. Signal Transduct Target Ther. 2023 Feb 24;8(1):76. doi: 10.1038/s41392-022-01286-3. PMID 36823150
- [Derived] Zhong WZ, Chen KN, Chen C, Gu CD, Wang J, Yang XN, Mao WM, Wang Q, Qiao GB, Cheng Y, Xu L, Wang CL, Chen MW, Kang X, Yan W, Yan HH, Liao RQ, Yang JJ, Zhang XC, Zhou Q, Wu YL. Erlotinib Versus Gemcitabine Plus Cisplatin as Neoadjuvant Treatment of Stage IIIA-N2 EGFR-Mutant Non-Small-Cell Lung Cancer (EMERGING-CTONG 1103): A Randomized Phase II Study. J Clin Oncol. 2019 Sep 1;37(25):2235-2245. doi: 10.1200/JCO.19.00075. Epub 2019 Jun 13. PMID 31194613
- See also: Induction Erlotinib Therapy in Stage III A (N2) Non-Small Cell Lung Cancer (NSCLC) — http://clinicaltrials.gov/ct2/show/NCT00600587